CLINICAL TRIAL: NCT07018024
Title: Prognosis of Anti-GBM Antibody Disease Through an International Cohort
Brief Title: Anti-Glomerular Basement Membrane Disease
Acronym: PRAGMATIC
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-05525-01
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-04

CONDITIONS: Anti-Glomerular Basement Membrane Disease
MeSH Terms: conditions — Anti-Glomerular Basement Membrane Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Plasma, serum and urine samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A: Patients diagnosed with anti-GBM disease 01-01-2010 until 31-12-2027 with available data about treatment
- Arm B: Patients diagnosed with anti-GBM disease, no time limit, with available blood and/or urine sample at time of diagnosis and information about if the patient was alive 6 months after treatment.

SUMMARY:
This study aims to clarify the prognosis of the rare but severe condition anti-glomerular basement membrane disease (anti-GBM disease also known as Goodpastures disease). Specifically, the aim is to investigate how the prognosis is affected by treatment options and disease severity at presentation measured using biomarkers in blood and urine. The study has two arms, one focusing on treatment (A) and one focusing on biomarkers (B). Data from a research subject (patient) can be included in both arms. For inclusion in arm A patients must be diagnosed after 01-01-2010 with available information about treatment and the participating clinic must have a search strategy enabling inclusion of > 80% of their patients. For inclusion in arm B there is no time limit, but there must be blood and/or urine samples available from the time of diagnosis and information about if the patient was alive six months after diagnosis.

Due to the rarity of anti-GBM disease, very few clinical trials have been conducted. Instead, available information comes from observational studies, most of which are relatively small and/or includes patients treated during the previous millennium, sometimes with sparse information about treatment. With this study we aim to collect more information about initial treatment. Today, treatment is based on three pharmaceutical groups; corticosteroids, cytotoxic agents and plasma exchange. Presently available data indicates that all three groups are needed, but all three can be used with variations in administration and intensity. At this time, it is not clear how intense the treatment needs to be, while it is clear that an intense treatment increases the risk of infections.

At present, two factors seem to be able to predict the possibility to preserve kidney function; kidney function at diagnosis measured as plasma creatinine concentration and the degree of kidney damage measured as the proportion of healthy renal corpuscles (glomeruli) in a tissue sample (biopsy). There is also data indicating that the amount of anti-GBM autoantibodies is prognostic, but this is less clear. In recent years, several other types of autoantibodies such as anti-laminin and anti-myeloperoxidase has been proposed to affect prognosis, but their importance remains unclear. Likewise, autoantibody characteristics such as subclass and exact binding site, can be evaluated, but the clinical significance of this is not known. This is also the case for markers of inflammation and renal damage in blood and urine.

ELIGIBILITY:
Arm A:

Inclusion Criteria:

* Anti-GBM disease diagnosed 01-01-2010 - 31-12-2027
* Available information about initial treatment

Arm B:

Inclusion Criteria:

* Anti-GBM disease diagnosis (no time limit)
* Available blood and/or urine sample at the time of diagnosis
* Available information about patient survival at six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for anti-GBM disease at one of the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Renal survival at 12 months | 12 months after diagnosis
  Measured as dialysis dependence

SECONDARY OUTCOMES:
Patient survival at six months | 6 months after diagnosis
Patient survival at 12 months | 12 months after diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Lund, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to the ethical regulations in Sweden. However, upon reasonable request to the study coordinators, selected anonymized data and/or data on group level might be shared.